CLINICAL TRIAL: NCT00098683
Title: A Phase II Study Of Amifostine In Children With Myelodysplastic Syndrome
Brief Title: Amifostine in Treating Young Patients With Newly Diagnosed De Novo Myelodysplastic Syndromes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: AAML0121; CDR0000398140 (Other: Clinical Trials.gov); COG-AAML0121 (Other: Children's Oncology Group)
Record Dates: First submitted 2004-12-07; First posted 2004-12-08 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: refractory anemia with excess blasts; refractory anemia; refractory anemia with ringed sideroblasts; de novo myelodysplastic syndromes; myelodysplastic/myeloproliferative neoplasm, unclassifiable; refractory cytopenia with multilineage dysplasia
MeSH Terms: conditions — Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Anemia, Refractory, with Excess of Blasts; Anemia, Refractory; Myeloproliferative Disorders | interventions — Amifostine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: amifostine trihydrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as amifostine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well amifostine works in treating young patients with newly diagnosed de novo myelodysplastic syndromes.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the hematologic effects of amifostine, in terms of, complete and partial response, in pediatric patients with newly diagnosed de novo myelodysplastic syndromes (MDS).
* Determine the safety and efficacy of this drug in these patients.

Secondary

* Determine the efficacy of this drug in preventing conversion of MDS to acute myeloid leukemia (AML) in terms of the proportion of patients who remain free of AML at the completion of study treatment.
* Determine the duration of progression-free remission from MDS conversion to AML in patients treated with this drug.
* Determine the effect of karyotypic abnormalities on survival and the duration from diagnosis of MDS until conversion to AML in patients treated with this drug.
* Determine the effect of bone marrow blast count on survival and the duration from diagnosis of MDS until conversion to AML in patients treated with this drug.
* Determine the effect of the number of cytopenias on survival in patients treated with this drug.
* Correlate the duration of time from diagnosis of MDS until conversion to AML with survival in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive amifostine IV over 1-3 minutes on days 1, 3, 5, 8, 10, 12, 15, 17, and 19. Treatment repeats every 5 weeks for 2 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease who are planning to undergo matched donor bone marrow or cord blood transplantation continue therapy until transplantation. Patients with stable or responding disease who are not undergoing transplantation may receive up to 4 additional courses of amifostine in the absence of disease progression or unacceptable toxicity.

Following completion of therapy with amifostine, patients are followed monthly for 1 year, every 2 months for 1 year, every 3 months for 1 year, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 10-20 patients will be accrued for this study within 5-10 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of myelodysplastic syndromes (MDS)

  * One of the following subtypes:

    * Refractory anemia (RA)
    * RA with ringed sideroblasts
    * RA with excess blasts
    * Refractory cytopenia with multilineage dysplasia (RCMD)
    * RCMD and ringed sideroblasts
    * MDS, unclassified
    * MDS associated with isolated del 5(q)
* De novo disease

  * No treatment-induced MDS
* No juvenile myelomonocytic leukemia
* No Down syndrome, Fanconi's anemia, or other inherited forms of hypoplastic bone marrow failure

PATIENT CHARACTERISTICS:

Age

* 1 to 21 at original diagnosis

Performance status

* Karnofsky 50-100% (patients > 16 years of age)
* Lansky 50-100% (patients 1 to 16 years of age)

Life expectancy

* At least 8 weeks

Hematopoietic

* See Disease Characteristics

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT < 2.5 times ULN

Renal

* Radioisotope glomerular filtration rate ≥ 60 mL/min OR
* Creatinine clearance > 60 mL/min (based on Schwartz formula)
* Calcium normal

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Serum electrolytes normal
* Phosphorus normal
* Magnesium normal
* Glucose normal
* No other concurrent malignancy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 8 weeks since prior growth factors
* No concurrent growth factors
* No concurrent hematopoietic stem cell transplantation
* No concurrent immunomodulating agents

Chemotherapy

* No prior amifostine
* No other concurrent anticancer chemotherapy

Endocrine therapy

* No concurrent daily steroid therapy

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No prior therapy for MDS

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2005-01; Primary Completion 2007-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Hematological effects (complete and partial response)
Safety and efficacy

SECONDARY OUTCOMES:
Efficacy
Duration of progression-free remission
Effect of karyotypic abnormalities on survival
Effect of the number of cytopenias on survival
Correlation of the duration of time from diagnosis of myelodysplastic syndromes until conversion to acute myeloid leukemia

CONTACTS AND LOCATIONS:
Overall Officials: Prasad Mathew, MD, Study Chair — University of New Mexico Cancer Center; Robert J. Arceci, MD, PhD — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (85):
- United States (74):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Long Beach, California
  - Children's Hospital Central California, Madera, California
  - Kaiser Permanente Medical Center - Oakland, Sacramento, California
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - Lee Cancer Care of Lee Memorial Health System, Fort Myers, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Miami Children's Hospital, Miami, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Kosair Children's Hospital, Louisville, Kentucky
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - CancerCare of Maine at Eastern Maine Medial Center, Bangor, Maine
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Spectrum Health Hospital - Butterworth Campus, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Overlook Hospital, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Maimonides Cancer Center at Maimonides Medical Center, Brooklyn, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Columbus Children's Hospital, Columbus, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Tod Children's Hospital - Forum Health, Youngstown, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Greenville Hospital System Cancer Center, Greenville, South Carolina
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine - Amarillo, Amarillo, Texas
  - Children's Hospital of Austin, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - West Virginia University - Robert C. Byrd Health Sciences Center - Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center at Cabell Huntington Hospital, Huntington, West Virginia
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (9):
  - University of Alberta Hospital, Edmonton, Alberta
  - Children's & Women's Hospital of British Columbia, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Montreal Children's Hospital at McGill University Health Center, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec
- San Jorge Children's Hospital, Santurce, Puerto Rico

REFERENCES:
- [Result] Mathew P, Gerbing R, Alonzo TA, Wallas T, Gong JZ, Jasty R, Jorstad DT, Raimondi SC, Chavez CM, Eisenberg NL, Hirsch B, Gamis A, Smith FO, Arceci RJ. A phase II study of amifostine in children with myelodysplastic syndrome: a report from the Children's Oncology Group study (AAML0121). Pediatr Blood Cancer. 2011 Dec 15;57(7):1230-2. doi: 10.1002/pbc.23164. Epub 2011 Jun 16. PMID 21681928